CLINICAL TRIAL: NCT03831737
Title: Team-based Ergonomics Educational Model for Workplace WELLNESS Improvement: A Pilot Study
Acronym: TEEM WELLNESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Aiesha Ahmed, Assistant Professor, Neuromuscular Neurology, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11328
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: MSDs; Muscle Pain
MeSH Terms: conditions — Myalgia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: In-Person (Experimental): During the initial 3 month control period, subjects are asked not to begin any new exercise or stretching program during this time.
  During the 3 month intervention period that follows, subjects will participate in in-person physical therapist-led instructional sessions three times per week. Each stretch will be performed twice, one on the left and one on the right. The therapist will describe what to do and briefly demonstrate each stretch. Stretches will be held for 45-60 seconds with therapist instructions and modification as needed based on subject technique.
  Interventions: Behavioral: stretching exercises
- Group 2: Video (Experimental): During the initial 3 month control period, subjects are asked not to begin any new exercise or stretching program during this time.
  During the 3 month intervention period that follows, subjects will complete sessions three times per week, led by a physical therapist and viewed remotely via pre-recorded video using a smartphone application.
  Interventions: Behavioral: stretching exercises

INTERVENTIONS:
Behavioral: stretching exercises — Head/neck stretches
  * Head tilt side to side
  * Cross-chest stretch Torso stretches
  * Side stretch
  * Mid-back stretch Lower limb
  * Standing quadriceps stretch
  * Standing hamstring stretch

SUMMARY:
This research is being done to explore the potential benefit of a physical therapist-guided stretching program on musculoskeletal pain and well-being.

ELIGIBILITY:
Inclusion Criteria:

* HMC/COM staff (faculty, residents, fellows, APPs, physical/occupational therapists, nurses, schedulers, etc.)
* At least 18 years old
* Willing and able to participate in all study procedures
* Willing and able to provide informed consent
* Group 2 subjects must have access to a computer with internet or an iPhone or Android smartphone

Exclusion Criteria:

* Subjects who do not meet all inclusion criteria will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
SF-36 | change from 3 month time point to 6 month time point
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.
CMDQ | change from 3 month time point to 6 month time point
  The Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) is a questionnaire based on previous published research studies of musculoskeletal discomfort among office workers.

SECONDARY OUTCOMES:
Modified Sit and Reach | baseline, 3 months, 6 months, change from 3 month time point to 6 month time point
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles.
SF-36 | baseline, 3 months
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.
CMDQ | baseline, 3 months
  The Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) is a questionnaire based on previous published research studies of musculoskeletal discomfort among office workers.

CONTACTS AND LOCATIONS:
Overall Officials: Aiesha Ahmed, MD, Principal Investigator — Penn State Health Milton S Hershey Medical Center; Majid Dadgar-Kiani, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No